CLINICAL TRIAL: NCT02502968
Title: A Double- Blind, Placebo Controlled, Randomized, Multicenter, Phase II Study to Assess the Efficacy of BL-8040 Addition to Consolidation Therapy in AML Patients
Brief Title: BL-8040 Addition to Consolidation Therapy in AML Patients
Acronym: BLAST
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Petra Tschanter (Other)
Collaborators: BioLineRx, Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Dr. Petra Tschanter, Dr. med., Martin-Luther-Universität Halle-Wittenberg
Organization: Martin-Luther-Universität Halle-Wittenberg (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UKH062014
Record Dates: First submitted 2015-07-06; First posted 2015-07-20 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; 4-fluorobenzoyl-TN-14003

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cytarabine & BL8040 (Experimental): Subjects ≥60 years: cytarabine 1g/m2 intravenously twice a day over 3 hours on day 1, 3 and 5 on 2 cycles and BL-8040 (1.25 mg/kg) subcutaneously on days 1 to 5 of each cycle
  Subjects <60 years: cytarabine 3g/m2 intravenously twice a day over 3 hours on day 1, 3 and 5 on 3 cycles and BL-8040 (1.25 mg/kg) subcutaneously on days 1 to 5 of each cycle
  Interventions: Drug: Cytarabine; Drug: BL-8040
- Cytarabine & Placebo (Active Comparator): Subjects ≥60 years: cytarabine 1g/m2 intravenously twice a day over 3 hours on day 1, 3 and 5 on 2 cycles and Placebo (for BL-8040) subcutaneously on days 1 to 5 of each cycle
  Subjects <60 years: cytarabine 3g/m2 intravenously twice a day over 3 hours on day 1, 3 and 5 on 3 cycles and Placebo (for BL-8040) subcutaneously on days 1 to 5 of each cycle
  Interventions: Drug: Cytarabine; Drug: Placebo (for BL-8040)

INTERVENTIONS:
Drug: Cytarabine
Drug: BL-8040
  Arms: Cytarabine & BL8040
Drug: Placebo (for BL-8040) — Powder for solution for injection manufactured to mimic BL-8040
  Arms: Cytarabine & Placebo

SUMMARY:
This study evaluates the addition of BL-8040 to the standard consolidation therapy with cytarabine in the treatment of acute myeloid leukemia (AML) in adults. Half of participants will receive BL-8040 and cytarabine in combination, while the other half will receive placebo and cytarabine.

DETAILED DESCRIPTION:
The majority of AML patients in first complete Remission (CR) do relapse despite the current consolidation therapy. Leukemic stem cells that are dormant in the bone marrow are presumed to be a major reason for AML relapse. Allogenic stem cell transplantation is an option only for a minority of AML patients in 1st CR. BL-8040 is a novel CXCR4 inhibitor that has a dual mechanism of action: inducing mobilization of leukemic blasts from the bone marrow which enhances cytotoxic effects of chemotherapy and has direct antileukemic, pro-apoptotic properties. The treatment with BL-8040 in combination with consolidation therapy (standard consolidation with high-dose cytarabine) should improve the efficacy of the consolidation therapy resulting in longer lasting remissions.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or morphologically confirmed diagnosis of AML except for AML M3 (acute promyelocytic leukemia)
* AML who achieved complete remission (CR), including CRi and CRp after a maximum number of 2 cycles of induction chemotherapy.
* AML subjects younger than 60 years at the time of diagnosis with intermediate or high-risk cytogenetics
* ECOG performance status ≤2
* Laboratory values as follows (at time of randomization): WBC < 30.000/μl and > 1000/μl, Platelets count > 70.000/μl, Creatinine < 1.0 mg/dl. If creatinine is between 1.0mg/dl and 1.3mg/dl, creatinine clearance should be > 30ml/min as calculated using the Cockroft-Gault formula
* Women of child-bearing potential must practice an acceptable method of birth control until 6 month after the last dose of treatment. Female subjects who are lactating must discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug.
* Male with a female partner of childbearing potential using a barrier method of contraception
* Written informed consent
* Subject is able and willing to comply with the requirements of the protocol.

Exclusion Criteria:

* Relapsed or refractory AML
* Start of induction cycle > 90 days before randomization.
* Subjects who have received >2 cycles of induction chemotherapy for AML therapy.
* Subjects younger than 60 years at the time of diagnosis with favorable cytogenetics (t(8;21) or inv(16) or t(16;16) or t(15;17)) or the confirmed presence of the resulting fusion protein AML1-ETO, CBFB-MYH11 or PML-RARA.
* Subjects for which allogeneic HSCT is planned in CR1.
* Planned further maintenance therapy after the end of the protocol defined consolidation therapy.
* Known allergic or hypersensitivity to BL8040- or cytarabine or to any of the test compounds, materials
* Use of investigational device or agents within 2 weeks or less than 5 half lifes for each investigational product /device at the time of enrolment. Registry studies are permissible.
* Abnormal liver function tests: Serum AST/ GOT or ALT/ GPT > 3x upper limit of normal (ULN), Serum bilirubin: Total bilirubin > 2.0mg/dl, conjugated bilirubin > 0.8mg/dl
* O2 saturation < 92% (on room air)
* Concurrent, uncontrolled medical condition, laboratory abnormality, or psychiatric illness which could place the subject at unacceptable risk
* Another malignancy within 3 years of enrolment, except in situ malignancy, or low-risk prostate, skin or cervical cancer after curative therapy. History of other cancer that according to the Investigator might confound the assessment of the endpoints of the study.
* A co-morbid condition which, in the view of the Investigators, renders the subject at high risk from treatment complications.
* History of any or more of the following cardiovascular conditions: cardiac angioplasty (within 6 months) or stenting (within 6 months) and/or myocardial infarction (MI) (within 6 months) or cerebro-vascular event within the past 6 months, unstable angina, vascular disease, class III or IV, congestive heart failure (as defined by the New York Heart Association (NYHA))
* Known central nervous system disease that may jeopardize the subject's study participation according to the investigator judgement
* Active, uncontrolled infection.
* Prior clinically significant grade 3-4 non-hematological toxicity to high-dose cytarabine or grade ≥ 2 of neurological toxicity
* Positive serology for HIV, active Hepatitis C and Hepatitis B (HBsAG pos.) at baseline
* Left ventricular ejection fraction (LVEF) of <40% by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO) at baseline
* Subjects with psychological, psychiatric, neurological, familial, sociological, or geographical conditions that do not permit compliance with the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Relapse Free Survival time | 18 months
  Relapse is defined as recurrence of leukemic blasts (more than 5%) in the bone marrow after confirmed complete remission

SECONDARY OUTCOMES:
Overall Survival | 18 months
Time to relapse | 18 months
Relapse free survival | 6, 9, 12 and 18 months
Relapse | 6, 9, 12 and 18 months
  Defined as recurrence of leukemic blasts (more than 5%) in the bone marrow after confirmed complete remission
Minimal residual disease | 6, 9, 12 and 18 months
  Immunophenotypic characterization of human bone marrow cells will be done to determine MRD
Toxicity | enitire study course until 18 months
  Number and CTC grade of all adverse events related to study treatment analyzed in an descriptive way

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Müller-Tidow, MD, Principal Investigator — University Hospital Halle, Germany
Locations (1):
- Univeritätsklinikum Halle, Klinik Innere Medizin 4, Halle, Germany